CLINICAL TRIAL: NCT03755596
Title: Clinical Evaluation of the Use of Ginger Extract in the Management of Motion Sickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação Educacional Serra dos Órgãos (Other)
Collaborators: Melora do Brasil Produtos Dermatológicos S/A (Unknown)
Responsible Party: Principal Investigator, Carlos Pereira Nunes, Principal Investigator, Fundação Educacional Serra dos Órgãos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOTC 01-05-18
Record Dates: First submitted 2018-11-23; First posted 2018-11-28 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Motion Sickness
Keywords: Zingiber officinale; Motion sickness; Motion sickness assessment questionnaire
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Intervention Model Description: Open-label, single-group, self-paired study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Oral treatment with single-dose 160mg Z. officinale extract in tablet form.
  Interventions: Drug: Z. officinale extract

INTERVENTIONS:
Drug: Z. officinale extract — Oral dose of 160mg dry ginger root (Z. officinale) extract in tablet form.

SUMMARY:
This is an open-label, case control study of 180 patients presenting motion sickness, who will perform a motion sickness assessment questionnaire before and after treatment with dry ginger (Z. officinale) extract.

DETAILED DESCRIPTION:
This open-label, self-paired, case-control study will evaluate 180 patients presenting motion sickness. The primary study objective is to evaluate the use of dry Z. officinale extract 160mg (containing 8mg gingerol) in the treatment of patients presenting motion sickness. The secondary objectives are to evaluate the effect of the treatment on the scores and subscores of the Motion Sickness Assessment Questionnaire (MSAQ) before and after treatment, as well as to assess treatment tolerability in this population. The total study duration will be seven days. A total of four specific motion sickness assessments will be performed, one pre-treatment and three during the treatment period, which consists of an oral dose of 160mg ginger extract 30 minutes prior to the trip under evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes between the ages of 18 and 65
* Clinical presentation of motion sickness
* Female participant of reproductive age agrees to use birth control during study period
* Patient has read, understood, signed and dated informed consent document

Exclusion Criteria:

* Hypersensitivity to any component of the study drug
* History of biliary calculus
* History of gastric irritation
* Hypertension > 145 / 100mmHg
* Concomitant use of other medicinal products for the treatment of motion sickness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
MSAQ total score change at Assessment 2 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change of 20 or more points on total MSAQ scores at Assessment 2 in relation to pretreatment scores.

SECONDARY OUTCOMES:
MSAQ total score change at Assessment 3 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change of 20 or more points on total MSAQ scores at Assessment 3 in relation to pretreatment scores.
MSAQ total score change at Assessment 4 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change of 20 or more points on total MSAQ scores at Assessment 4 in relation to pretreatment scores.
MSAQ subscore change at Assessment 2 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change on MSAQ subscores at Assessment 2 in relation to pretreatment scores.
MSAQ subscore change at Assessment 3 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change on MSAQ subscores at Assessment 3 in relation to pretreatment scores.
MSAQ subscore change at Assessment 4 | MSAQ completed within 30 minutes of car, bus, boat, ferry, or train ride lasting at least 15 minutes.
  Percentage of patients presenting change on MSAQ subscores at Assessment 4 in relation to pretreatment scores.
Adverse event occurrence | From first dose to end of study (no more than 7 days from Pretreatment visit date)
  Number of subjects reporting adverse effects during treatment period

OTHER OUTCOMES:
Physician Assessment score change | Scores taken at pretreatment and at the end of the treatment period (no more than 7 days).
  Mean Physician Assessment (10-point scale assessing overall patient condition ranging from 1 [worst] to 10 [best]) score improvement at end-of-study visit compared to pretreatment scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário Serra dos Órgãos - UNIFESO, Teresópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No